CLINICAL TRIAL: NCT00529880
Title: Fludarabine and Cytarabine as Continuous Infusion Plus G-CSF Priming for Elderly Patients With Resistant AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-008
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2007-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fludarabine , cytarabine

SUMMARY:
* To determine the feasibility of fludarabine and cytarabine as continuous infusion plus granulocyte-colony stimulating factor priming for elderly patients with resistant acute myeloid leukemia other than acute promyelocytic leukemia
* The feasibility will be evaluated in terms of toxicities, complete remission rate, duration of complete remission, disease-free survival, and overall survival.

DETAILED DESCRIPTION:
* A second course of induction chemotherapy can be given to the patient when a partial remission but less than a complete remission is achieved after the first course. At least 4 weeks should be apart between start of the first course and start of the second course.
* G-CSF (Lenograstim) 250 g/day will begin to be administered after the confirmation of hypocellular bone marrow with blasts less than 5% on day 14 or later until absolute neutrophil counts are 1,000/l or more.
* For the patients who achieve a complete remission, consolidation therapy will be given as follows:

  * Two more cycles of the same chemotherapy will be given to the patients who achieve a complete remission after single induction course. Allogeneic or autologous hematopoietic cell transplantation could be also considered.
  * In patients who relapse after allogeneic hematopoietic cell transplantation, donor leukocyte infusion will be done without consolidation chemotherapy.
  * In patients who had extramedullary relapse(s), local radiotherapy can be given to the relapse site(s).

ELIGIBILITY:
Inclusion Criteria:

* Failure to achieve CR after initial induction chemotherapy
* Any relapse, regardless of the frequency and time of relapse from first CR
* Relapse after hematopoietic cell transplantation, allogeneic or autologous.
* Multiple relapses, extramedullary relapse(s)

Exclusion Criteria:

* Inadequate hepatic,renal,cardiac function
* Psychiatric disorder or mental deficiency
* CNS involvement of leukemic blasts

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2004-12; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate, duration of complete remission, toxicities

SECONDARY OUTCOMES:
progression-free survival, overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hawk Kim, professor, Principal Investigator — Ulsan University Hospital, ROK
Locations (1):
- Asan Medical Center, Songpa-gu, Seoul, South Korea